CLINICAL TRIAL: NCT04574947
Title: Intravenous Or Topical Lidocaine And Neuromonitoring in Thyroid Surgery (IOLANT Study)
Brief Title: Lidocaine And Neuromonitoring in Thyroid Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Saint Petersburg State University, Russia (Other)
Responsible Party: Principal Investigator, Efremov Sergey, Principal investigator, Saint Petersburg State University, Russia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IOLANT
Record Dates: First submitted 2020-09-24; First posted 2020-10-05 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Thyroid Neoplasm; Parathyroid Neoplasms; Anesthesia
MeSH Terms: conditions — Thyroid Neoplasms; Parathyroid Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intravenous lidocaine (Active Comparator)
  Interventions: Drug: Intravenous lidocaine; Procedure: Intra-cuff placebo
- Topical lidocaine (Experimental)
  Interventions: Drug: Intravenous placebo; Procedure: Intra-cuff lidocaine
- Placebo (Placebo Comparator)
  Interventions: Drug: Intravenous placebo; Procedure: Intra-cuff placebo

INTERVENTIONS:
Drug: Intravenous lidocaine — Lidocaine IV 1.5 mg / kg BMI will be administered during induction into anaesthesia followed by infusion at a dose of 1.5 mg / kg / h until the end of the surgery.
  Arms: Intravenous lidocaine
Drug: Intravenous placebo — During induction and maintenance of anaesthesia, 0.9% sodium chloride solution will be injected intravenously at a rate equivalent to lidocaine solution.
  Arms: Placebo; Topical lidocaine
Procedure: Intra-cuff lidocaine — The lidocaine solution will be applied to the intubation tube and the cuff will be filled with an alkalinised lidocaine solution.
  Arms: Topical lidocaine
Procedure: Intra-cuff placebo — The intubation tube will be lubricated 0.9% sodium chloride, the tube cuff will be filled with 0.9% sodium chloride solution.
  Arms: Intravenous lidocaine; Placebo

SUMMARY:
The aim of this study is to test the hypothesis that the quality of recovery with topical lidocaine is better than placebo.

DETAILED DESCRIPTION:
The use of neuromonitoring in thyroid surgery imposes a number of special demands for anaesthetic management. Such demands include avoiding muscle relaxation and local anaesthesia. Maintaining a balance between the risk of awakening during surgery and excessively deep anaesthesia in fast track surgery is an important task for the anaesthesiologist.

Mild anaesthesia in the absence of muscle relaxation increases the risk of developing laryngeal reflexes, coughing during surgery, while excessively deep anaesthesia slows down recovery after surgery and increases the risk of arterial hypotension. The frequency and duration of arterial hypotension, as well as the depth of anesthesia assessed by the Bispectral index, are independent risk factors for postoperative cardiovascular complications and long-term mortality. On the other hand, coughing in response to irritation of the endotracheal tube during recovery from anesthesia is recognized as a risk factor for respiratory and cardiovascular complications, as well as postoperative wound insufficiency.

Optimization the anesthesia by intravenous infusion of lidocaine can improve anesthesia controllability, hemodynamic stability and overall anesthesia recovery rates. Local use of lidocaine, including filling the endotracheal tube cuff with its alkalinized solution, has also been shown to be effective in reducing the frequency of laryngeal reflexes upon awakening after surgery of varying duration. However, the efficacy and safety of local use of lidocaine under neuromonitoring conditions has not been studied. Despite recommendations to avoid the local use of lidocaine for tracheal intubation, there is evidence of the safety of this technique in the absence of a negative impact on the quality of neuromonitoring.

The purpose of this study is to test the hypothesis that the quality of recovery with topical lidocaine is better than placebo. At the same time, the investigators assume that recovery after surgery will be comparable with both local and intravenous use. Intergroup differences in arterial hypotension, depth of anesthesia and intraoperative neuromonitoring parameters will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Planned thyroid surgery
* Age> 45 years
* Signed informed consent to participate in the study

Exclusion Criteria:

* Emergency surgery
* Redo surgery
* Contraindications for lidocaine use
* Pregnancy
* Enrolment to another randomised clinical trial within the last 30 days

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Quality of recovery 40 questionnaire | First postoperative day
  Minimum and maximum values: 40 and 200, where higher scores mean a better outcomes

SECONDARY OUTCOMES:
Hypotension incidence | Intraoperative
  Incidence of arterial hypotension (SBP <60 mm Hg)
Hypotension duration | Intraoperative
  Cumulative duration of arterial hypotension (SBP <60 mm Hg) expressed in minutes
Cough rate | In the operating room and during awakening.
  Frequency of laryngeal reflexes
Minimal bispectral index | During surgery
  Minimal observed intraoperative bispectral index value. Values less than 40 mean a worse outcomes.
Bispectral index less then 40 | During surgery
  Cumulative duration of bispectral index less than 40. Values less than 40 mean a worse outcomes.
Amplitude | During surgery
  Amplitude of electromyographic potential during neuromonitoring of recurrent nerve
Latency | During surgery
  Latency of electromyographic potential during neuromonitoring of recurrent nerve

CONTACTS AND LOCATIONS:
Locations (1):
- St. Petersburg State University Hospital, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code